CLINICAL TRIAL: NCT04605289
Title: Biochemical Efficacy of Cymbopogon Citratus Gel as Local Drug Delivery Agent in Reducing Matrix Metalloproteinase-8 Levels Intra-crevicularly in Moderate Periodontitis Patients
Brief Title: Levels of Matrix Metalloproteinase-8 After Intrapocket Treatment in Moderate Periodontitis Patients.
Acronym: MMP-8
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Nadein El Sharif, A student of Master's degree, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17102019
Record Dates: First submitted 2020-10-15; First posted 2020-10-28 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Intervention Model Description: -Cymbopogon citratus oil gel /-Placebo gel. will be intrapocket application as an adjunctive treatment to conventional therapy
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (study group) (Experimental): Scaling and root planing + intra-pocket application of 2% Cymbopogon citratus (lemon-grass) gel
  Interventions: Drug: lemongrass essential oil gel; Procedure: Scaling and root planing
- Group II (control group) (Placebo Comparator): Scaling and root planing +intra-pocket application of placebo gel
  Interventions: Drug: Placebo; Procedure: Scaling and root planing

INTERVENTIONS:
Drug: lemongrass essential oil gel — The lemongrass oil gel will be administered by means of a syringe with a bent, blunt-end needle. The needle will be carefully inserted into the periodontal pocket and the gel will be applied in the test sites in a gentle probing manner, attempting to fill the full extent of the pocket. The gel will be applied up to the gingival margin and the excess gel will be removed with sterile gauze.
  Periodontal dressing will be applied after the delivery of the drug, and they will be also asked not to eat for thirty minutes.
  After placement of the gel in situ, patients will be instructed to follow strict oral hygiene protocol and not chew hard or sticky foods at the gel placement sites for rest of the week.
  Other Names: Cymbopogon citratus oil gel
  Arms: Group I (study group)
Drug: Placebo — The placebo will be administered by means of a syringe with a bent, blunt-end needle. The needle will be carefully inserted into the periodontal pocket and the gel will be applied in the test sites in a gentle probing manner, attempting to fill the full extent of the pocket. The gel will be applied up to the gingival margin and the excess gel will be removed with sterile gauze.
  Periodontal dressing will be applied after the delivery of the drug, and they will be also asked not to eat for thirty minutes.
  After placement of the gel in situ, patients will be instructed to follow strict oral hygiene protocol and not chew hard or sticky foods at the gel placement sites for rest of the week.
  Other Names: Carbopol®-Based pH-Sensitive gel
  Arms: Group II (control group)
Procedure: Scaling and root planing — Conventional mechanical treatment by ultra-sonic scalers

SUMMARY:
Using local delivery drugs as adjunctive to scaling and root planing and evaluating gingival crevicular fluid (GCF) biological molecular markers (MMP-8).

DETAILED DESCRIPTION:
Study sample and setting A sample size of twenty patients per group (number of groups = 2) (total sample size = 40 patients) is the sufficient required sample as statistically significant with 80% power. The sample size was calculated using g power version 3.1.9.2. patients will be recruited from the outpatient clinic of the Department of Oral Medicine, Periodontology, Diagnosis and Oral Radiology. Faculty of Dentistry, Alexandria University.

Treatment will be in accordance with the principles of the modified Helsinki code for human clinical studies (2013).

The clinical study will be conducted following the ethical guidelines for conduct of research on human subjects, by the Faculty of Dentistry, Alexandria University (IRB NO:00010556 - IORG 0008839).

Data management and statistical analysis The data will be processed and analysed using statistical package for social sciences program SPSS (20.0) software*. The study will include descriptive and analytical data. A P-value of less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes having moderate periodontitis (stage II), CAL 3-4mm.
2. Patients' age between 25 and 45 years old.
3. Systemically healthy patients.
4. No history of periodontal therapy (surgical and non-surgical) or taken any antibiotic therapy for the past six months.

Exclusion Criteria:

1. History of smoking.
2. Patients having previous adverse reaction to the products (or similar products) used in this study.
3. Grade C category that has rapid rate of progression.
4. Pregnant and lactating women.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
Changes of clinical attachment and periodontal probing pocket | at baseline and twelve weeks from intervention.
  Millimeters (mm)

SECONDARY OUTCOMES:
GCF concentration of MMP-8 | at baseline, one week, and twelve weeks from intervention.
  pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Nadein E Sharif, Principal Investigator — Alexandria University
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Bascones-Martinez A, Munoz-Corcuera M, Noronha S, Mota P, Bascones-Ilundain C, Campo-Trapero J. Host defence mechanisms against bacterial aggression in periodontal disease: Basic mechanisms. Med Oral Patol Oral Cir Bucal. 2009 Dec 1;14(12):e680-5. doi: 10.4317/medoral.14.e680. PMID 19680192
- [Background] Preshaw M. Periodontal disease pathogenesis. 13th ed. Newman M, Takei H, Klokkevold P, Carranza F, editors. Philadelphia: Elsevier - Health Sciences Division; 2018.
- [Background] Caton JG, Armitage G, Berglundh T, Chapple ILC, Jepsen S, Kornman KS, Mealey BL, Papapanou PN, Sanz M, Tonetti MS. A new classification scheme for periodontal and peri-implant diseases and conditions - Introduction and key changes from the 1999 classification. J Clin Periodontol. 2018 Jun;45 Suppl 20:S1-S8. doi: 10.1111/jcpe.12935. PMID 29926489
- [Background] Tonetti MS, Greenwell H, Kornman KS. Staging and grading of periodontitis: Framework and proposal of a new classification and case definition. J Clin Periodontol. 2018 Jun;45 Suppl 20:S149-S161. doi: 10.1111/jcpe.12945. PMID 29926495
- [Background] Needleman I, Garcia R, Gkranias N, Kirkwood KL, Kocher T, Iorio AD, Moreno F, Petrie A. Mean annual attachment, bone level, and tooth loss: A systematic review. J Clin Periodontol. 2018 Jun;45 Suppl 20:S112-S129. doi: 10.1111/jcpe.12943. PMID 29926483
- [Background] Taba M Jr, Kinney J, Kim AS, Giannobile WV. Diagnostic biomarkers for oral and periodontal diseases. Dent Clin North Am. 2005 Jul;49(3):551-71, vi. doi: 10.1016/j.cden.2005.03.009. PMID 15978241
- [Background] Hernández-Ríos P, Hernández M, Garrido M, Tervahartiala T, Leppilahti J, Kuula H, et al. Oral fluid matrix metalloproteinase (MMP)-8 as a diagnostic tool in chronic periodontitis. Dove Press. 2016; 2016(30):11-18.
- [Background] Goodson JM. Diagnosis of Periodontitis by Physical Measurement: Interpretation From Episodic Disease Hypothesis. J Periodontol. 1992 Apr;63 Suppl 4S:373-382. doi: 10.1902/jop.1992.63.4s.373. PMID 29539683
- [Background] Griffiths GS. Formation, collection and significance of gingival crevice fluid. Periodontol 2000. 2003;31:32-42. doi: 10.1034/j.1600-0757.2003.03103.x. No abstract available. PMID 12656994
- [Background] Kinney JS, Morelli T, Braun T, Ramseier CA, Herr AE, Sugai JV, Shelburne CE, Rayburn LA, Singh AK, Giannobile WV. Saliva/pathogen biomarker signatures and periodontal disease progression. J Dent Res. 2011 Jun;90(6):752-8. doi: 10.1177/0022034511399908. Epub 2011 Mar 15. PMID 21406610
- [Background] Kinney JS, Morelli T, Oh M, Braun TM, Ramseier CA, Sugai JV, Giannobile WV. Crevicular fluid biomarkers and periodontal disease progression. J Clin Periodontol. 2014 Feb;41(2):113-120. doi: 10.1111/jcpe.12194. Epub 2013 Dec 12. PMID 24303954
- [Background] Wilton JM, Curtis MA, Gillett IR, Griffiths GS, Maiden MF, Sterne JA, Wilson DT, Johnson NW. Detection of high-risk groups and individuals for periodontal diseases: laboratory markers from analysis of saliva. J Clin Periodontol. 1989 Sep;16(8):475-83. doi: 10.1111/j.1600-051x.1989.tb02323.x. PMID 2674204
- [Background] Srivastava N, Nayak PA, Rana S. Point of Care- A Novel Approach to Periodontal Diagnosis-A Review. J Clin Diagn Res. 2017 Aug;11(8):ZE01-ZE06. doi: 10.7860/JCDR/2017/26626.10411. Epub 2017 Aug 1. PMID 28969294
- [Background] Teles RP, Haffajee AD, Socransky SS. Microbiological goals of periodontal therapy. Periodontol 2000. 2006;42:180-218. doi: 10.1111/j.1600-0757.2006.00192.x. No abstract available. PMID 16930311
- [Background] Aimetti M. Nonsurgical periodontal treatment. Int J Esthet Dent. 2014 Summer;9(2):251-67. PMID 24765632
- [Background] Zandbergen D, Slot DE, Cobb CM, Van der Weijden FA. The clinical effect of scaling and root planing and the concomitant administration of systemic amoxicillin and metronidazole: a systematic review. J Periodontol. 2013 Mar;84(3):332-51. doi: 10.1902/jop.2012.120040. Epub 2012 May 21. PMID 22612369
- [Background] Tariq M, Iqbal Z, Ali J, Baboota S, Talegaonkar S, Ahmad Z, Sahni JK. Treatment modalities and evaluation models for periodontitis. Int J Pharm Investig. 2012 Jul;2(3):106-22. doi: 10.4103/2230-973X.104394. PMID 23373002
- [Background] Sethi K, Kale A, Mahale S, Karde P, Mamajiwala A, Sonawane S. Comparative evaluation of clinical and microbiological efficacy of 2% lemongrass gel versus 1%chlorhexidine gel as a local drug delivery system in the treatment of chronic periodontitis: a randomized controlled clinical trial. Int J Adv Res. 2018; 6(7):381-388.
- [Background] Moro MG, Silveira Souto ML, Franco GCN, Holzhausen M, Pannuti CM. Efficacy of local phytotherapy in the nonsurgical treatment of periodontal disease: A systematic review. J Periodontal Res. 2018 Jun;53(3):288-297. doi: 10.1111/jre.12525. Epub 2018 Jan 19. PMID 29352465
- [Background] Bhat G, Kudva P, Dodwad V. Aloe vera: Nature's soothing healer to periodontal disease. J Indian Soc Periodontol. 2011 Jul;15(3):205-9. doi: 10.4103/0972-124X.85661. PMID 22028505
- [Background] Grover S, Tewari S, Sharma RK, Singh G, Yadav A, Naula SC. Effect of Subgingivally Delivered 10% Emblica officinalis Gel as an Adjunct to Scaling and Root Planing in the Treatment of Chronic Periodontitis - A Randomized Placebo-controlled Clinical Trial. Phytother Res. 2016 Jun;30(6):956-62. doi: 10.1002/ptr.5600. Epub 2016 Feb 24. PMID 26914986
- [Background] Phogat M, Rana T, Prasad N, Baiju CS. Comparative evaluation of subgingivally delivered xanthan-based chlorhexidine gel and herbal extract gel in the treatment of chronic periodontitis. J Indian Soc Periodontol. 2014 Mar;18(2):172-7. doi: 10.4103/0972-124X.131319. PMID 24872624
- [Background] Warad SB, Kolar SS, Kalburgi V, Kalburgi NB. Lemongrass essential oil gel as a local drug delivery agent for the treatment of periodontitis. Anc Sci Life. 2013 Apr;32(4):205-11. doi: 10.4103/0257-7941.131973. PMID 24991068
- [Background] Jayasinha P. Lemongrass. In. Colombo: Industrial Technology Institute; 1999. 1-45.
- [Background] Souza Formigoni ML, Lodder HM, Gianotti Filho O, Ferreira TM, Carlini EA. Pharmacology of lemongrass (Cymbopogon citratus Stapf). II. Effects of daily two month administration in male and female rats and in offspring exposed "in utero". J Ethnopharmacol. 1986 Jul;17(1):65-74. doi: 10.1016/0378-8741(86)90073-5. PMID 3762196
- [Background] Leite JR, Seabra Mde L, Maluf E, Assolant K, Suchecki D, Tufik S, Klepacz S, Calil HM, Carlini EA. Pharmacology of lemongrass (Cymbopogon citratus Stapf). III. Assessment of eventual toxic, hypnotic and anxiolytic effects on humans. J Ethnopharmacol. 1986 Jul;17(1):75-83. doi: 10.1016/0378-8741(86)90074-7. PMID 2429120
- [Background] Choudhury S. Effect of clipping height on herb and essential oil yield of Cymbopogon. Indian J Agron. 1994;39(4):592-598
- [Background] Manvitha K, Bidya B. Review on pharmacological activity of cymbopogon citratus. Int. J. Herb. Med. 2014;1(6): 5-7.
- [Background] Mulyaningsih S, Sporer F, Reichling J, Wink M. Antibacterial activity of essential oils from Eucalyptus and of selected components against multidrug-resistant bacterial pathogens. Pharm Biol. 2011 Sep;49(9):893-9. doi: 10.3109/13880209.2011.553625. Epub 2011 May 19. PMID 21591991
- [Background] Sadlon AE, Lamson DW. Immune-modifying and antimicrobial effects of Eucalyptus oil and simple inhalation devices. Altern Med Rev. 2010 Apr;15(1):33-47. PMID 20359267
- [Background] Ghosh G. Traditional use of plants against leprosy in India: a review of the recent literature. J Innov Pharm Biol Sci. 2017;4(4): 55-64.
- [Background] Silva-Neto RP, Peres MF, Valenca MM. Odorant substances that trigger headaches in migraine patients. Cephalalgia. 2014 Jan;34(1):14-21. doi: 10.1177/0333102413495969. Epub 2013 Jul 5. PMID 23832131
- [Background] Arrey Tarkang P, Franzoi KD, Lee S, Lee E, Vivarelli D, Freitas-Junior L, Liuzzi M, Nole T, Ayong LS, Agbor GA, Okalebo FA, Guantai AN. In vitro antiplasmodial activities and synergistic combinations of differential solvent extracts of the polyherbal product, Nefang. Biomed Res Int. 2014;2014:835013. doi: 10.1155/2014/835013. Epub 2014 Apr 27. PMID 24877138
- [Background] Arrey Tarkang P, Nwachiban Atchan AP, Kuiate JR, Okalebo FA, Guantai AN, Agbor GA. Antioxidant potential of a polyherbal antimalarial as an indicator of its therapeutic value. Adv Pharmacol Sci. 2013;2013:678458. doi: 10.1155/2013/678458. Epub 2013 Dec 19. PMID 24454347
- [Background] Figueirinha A, Francisco V, Costa G, Liberal J, Lopes M, García-Rodríguez C, et al. Chemical characterization and anti-inflammatory activity of luteolin glycosides isolated from lemongrass. J Funct Foods. 2014;10(2):436-443
- [Background] Francisco V, Costa G, Figueirinha A, Marques C, Pereira P, Miguel Neves B, Celeste Lopes M, Garcia-Rodriguez C, Teresa Cruz M, Teresa Batista M. Anti-inflammatory activity of Cymbopogon citratus leaves infusion via proteasome and nuclear factor-kappaB pathway inhibition: contribution of chlorogenic acid. J Ethnopharmacol. 2013 Jun 21;148(1):126-34. doi: 10.1016/j.jep.2013.03.077. Epub 2013 Apr 10. PMID 23583902
- [Background] Meenapriya M, Priya J. Effects of lemongrass oil on rheumatoid arthritis. J Pharm Sci & Res. 2017;9(2): 237-239.
- [Background] de Cassia da Silveira e Sa R, Andrade LN, de Sousa DP. A review on anti-inflammatory activity of monoterpenes. Molecules. 2013 Jan 18;18(1):1227-54. doi: 10.3390/molecules18011227. PMID 23334570
- [Background] Anand M, Goyal R, Bhat S, Kamath S, Aggarwal M, Bhandarkar M, et al. A novel anti-oxidant lemon grass oil mouth wash-a clinical trial. J Exp Biol Sci. 2011;2(3): 59-64.
- [Background] Kumar S, Gurunathan D. Lemongrass in dental health. Drug Invention Today. 2019;11(3): 780-785.
- [Background] Prabahar C, Nivetha R. Evaluation of efficacy of lemongrass gel as a local drug delivery with chlorhexidine gel in chronic periodontitis -a comparative study. Int J Adv Res. 2017;6(9): 6017-6020.
- [Background] Kumar S, Himmelstein KJ. Modification of in situ gelling behavior of carbopol solutions by hydroxypropyl methylcellulose. J Pharm Sci. 1995 Mar;84(3):344-8. doi: 10.1002/jps.2600840315. PMID 7616375
- [Background] Gul SS, Griffiths GS, Stafford GP, Al-Zubidi MI, Rawlinson A, Douglas CWI. Investigation of a Novel Predictive Biomarker Profile for the Outcome of Periodontal Treatment. J Periodontol. 2017 Nov;88(11):1135-1144. doi: 10.1902/jop.2017.170187. Epub 2017 Jul 3. PMID 28671508
- [Background] Nedzi-Gora M, Gorska R, Kostrzewa-Janicka J, Kowalski J. Concentration of MMP-8 and IL-1beta in gingival crevicular fluid in patients with chronic and aggressive periodontitis. Cent Eur J Immunol. 2017;42(4):342-346. doi: 10.5114/ceji.2017.72824. Epub 2017 Dec 30. PMID 29472810
- [Background] Buduneli N, Kinane DF. Host-derived diagnostic markers related to soft tissue destruction and bone degradation in periodontitis. J Clin Periodontol. 2011 Mar;38 Suppl 11:85-105. doi: 10.1111/j.1600-051X.2010.01670.x. PMID 21323706
- [Background] Sorsa T, Tjaderhane L, Salo T. Matrix metalloproteinases (MMPs) in oral diseases. Oral Dis. 2004 Nov;10(6):311-8. doi: 10.1111/j.1601-0825.2004.01038.x. PMID 15533204
- [Background] Reinhardt RA, Stoner JA, Golub LM, Lee HM, Nummikoski PV, Sorsa T, Payne JB. Association of gingival crevicular fluid biomarkers during periodontal maintenance with subsequent progressive periodontitis. J Periodontol. 2010 Feb;81(2):251-9. doi: 10.1902/jop.2009.090374. PMID 20151804
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c869. doi: 10.1136/bmj.c869. No abstract available. PMID 20332511
- [Background] Christodoulides N, Nikolidakis D, Chondros P, Becker J, Schwarz F, Rossler R, Sculean A. Photodynamic therapy as an adjunct to non-surgical periodontal treatment: a randomized, controlled clinical trial. J Periodontol. 2008 Sep;79(9):1638-44. doi: 10.1902/jop.2008.070652. PMID 18771363
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Ismail FA, Napaporn J, Hughes JA, Brazeau GA. In situ gel formulations for gene delivery: release and myotoxicity studies. Pharm Dev Technol. 2000;5(3):391-7. doi: 10.1081/pdt-100100555. PMID 10934739
- [Background] Kim J, Shin W. How to do random allocation (randomization). Clin Orthop Surg. 2014 Mar;6(1):103-9. doi: 10.4055/cios.2014.6.1.103. Epub 2014 Feb 14. PMID 24605197
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c332. doi: 10.1136/bmj.c332. PMID 20332509
- [Background] Lenox JA, Kopczyk RA. A clinical system for scoring a patient's oral hygiene performance. J Am Dent Assoc. 1973 Apr;86(4):849-52. doi: 10.14219/jada.archive.1973.0178. No abstract available. PMID 4511175
- [Background] Glavind L, Loe H. Errors in the clinical assessment of periodontal destruction. J Periodontal Res. 1967;2(3):180-4. doi: 10.1111/j.1600-0765.1967.tb01887.x. No abstract available. PMID 4237475
- [Background] Loe H. The Gingival Index, the Plaque Index and the Retention Index Systems. J Periodontol. 1967 Nov-Dec;38(6):Suppl:610-6. doi: 10.1902/jop.1967.38.6.610. No abstract available. PMID 5237684
- [Background] Azouni KG, Tarakji B. The trimeric model: a new model of periodontal treatment planning. J Clin Diagn Res. 2014 Jul;8(7):ZE17-20. doi: 10.7860/JCDR/2014/8458.4623. Epub 2014 Jul 20. PMID 25177662
- [Background] Do J, Takei H, Carranza F. The Treatment Plan. In Newman M, Takei H, Klokkevold P, Carranza F. Newman and Carranza's Clinical Periodontology. 13th ed. Philadelphia: Elsevier - Health Sciences Division; 2018. 426-430.
- [Background] Goodson J. Intra-pocket drug delivery devices for treatment of periodontal. U.S. Patent. 1988.
- [Background] Guentsch A, Kramesberger M, Sroka A, Pfister W, Potempa J, Eick S. Comparison of gingival crevicular fluid sampling methods in patients with severe chronic periodontitis. J Periodontol. 2011 Jul;82(7):1051-60. doi: 10.1902/jop.2011.100565. Epub 2011 Jan 14. PMID 21235330
- [Background] Kinane DF, Darby IB, Said S, Luoto H, Sorsa T, Tikanoja S, Mantyla P. Changes in gingival crevicular fluid matrix metalloproteinase-8 levels during periodontal treatment and maintenance. J Periodontal Res. 2003 Aug;38(4):400-4. doi: 10.1034/j.1600-0765.2003.00663.x. PMID 12828657
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2019-10-17): https://cdn.clinicaltrials.gov/large-docs/89/NCT04605289/Prot_ICF_000.pdf